CLINICAL TRIAL: NCT03268681
Title: BIOtinidase Test In Optic-Neuropathy
Acronym: BIOTIN
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RDS_2017_14
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Biotin Deficiency; Optic Neuropathy
MeSH Terms: conditions — Biotin deficiency; Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biotinidase is an enzyme that recycles biotin, a water-soluble vitamin essential as a coenzyme for four carboxylases that are involved in gluconeogenesis, fatty acid synthesis, and in the catabolism of several branch-chain amino acids. Biotinidase deficiency (BD) is an autosomal recessively inherited disorder. Patients with profound BD (<10% of mean normal serum biotinidase activity) presents, usually during early childhood, with neurological (seizures, hypotonia, ataxia, developmental delay, vision problems, and/or hearing loss) and non-neurological findings (metabolic acidosis, respiratory difficulties, alopecia and/or skin rash) that may progress to coma or death if untreated.

Three cases of adult-onset biotinidase deficiency with reversible optic neuropathy have recently been described in France, where there is no neonatal screening of BP. Once treated with Biotin, patients' vision was fully restored.

This study aims to assess the prevalence of BP among a population of patients with idiopathic optic neuropathy, and to assess the efficacy of Biotin supplementation on visual impairment in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with bilateral optic neuropathy
* symptoms beginning before 50 years old
* diagnosed for more than 1 months
* etiology unknown

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopatic bilateral optic neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
prevalence of biotin deficiency among patients with idiopathic optic neuropathy | baseline
  measure of biotinidase activity (nkat/l unit)

CONTACTS AND LOCATIONS:
Overall Officials: Romain Deschamps, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation OPH A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No